CLINICAL TRIAL: NCT02624388
Title: A Randomized, Placebo-Controlled Pilot Study of Genistein Supplementation in Pediatric Cancer Patients Receiving Myelosuppressive Chemotherapy
Brief Title: Study of Genistein in Pediatric Oncology Patients (UVA-Gen001)
Acronym: UVA-Gen001
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: Poor enrollment
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, William Petersen, MD, Director, Pediatric Novel Therapeutics Program (Hematology/Oncology), University of Virginia
Allocation: Randomized | Model: Crossover | Masking: Triple | Purpose: Supportive Care
Other Study IDs: 17588
Record Dates: First submitted 2015-10-27; First posted 2015-12-08 (Estimated); Results first posted 2024-05-06 (Actual); Last update posted 2024-05-06 (Actual); Status verified 2024-05

CONDITIONS: Lymphoma; Childhood Lymphoma; Solid Tumor; Childhood Solid Tumor; Neuroblastoma; Ewing Sarcoma; Hodgkin Lymphoma; Non-Hodgkin Lymphoma; Rhabdomyosarcoma; Soft Tissue Sarcoma; Medulloblastoma; Germ Cell Tumor; Wilms Tumor; Brain Neoplasms; Medulloblastoma, Childhood; Neuroectodermal Tumors, Primitive
Keywords: Genistein; Soy; Chemotherapy side-effects; Pediatric Cancer; Isoflavone
MeSH Terms: conditions — Lymphoma; Neuroblastoma; Sarcoma, Ewing; Hodgkin Disease; Lymphoma, Non-Hodgkin; Rhabdomyosarcoma; Sarcoma; Medulloblastoma; Neoplasms, Germ Cell and Embryonal; Wilms Tumor; Brain Neoplasms; Neuroectodermal Tumors, Primitive; Neoplasms | interventions — Genistein

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Arm A: Genistein followed by Placebo (Experimental): Genistein daily throughout chemotherapy cycles 1 and 2, and placebo daily during chemotherapy cycles 3 and 4
  Interventions: Drug: Genistein; Drug: Placebo
- Arm B: Placebo followed by Genistein (Experimental): Placebo daily throughout chemotherapy cycles 1 and 2, and genistein daily during chemotherapy cycles 3 and 4
  Interventions: Drug: Genistein; Drug: Placebo

INTERVENTIONS:
Drug: Genistein — Estrogen-like compound (isoflavone) derived from soybeans
  Other Names: 5, 7-dihydroxy-3-(4-hydroxyphenyl)-4H-1-benzopyran-4-one; i-cool tablets containing 30 mg geniVida™
Drug: Placebo — Pill that contains no medicine

SUMMARY:
Toxicities related to pediatric cancer treatment can lead to significant illness, organ damage, treatment delays, increased health care cost, and decrease in quality of life. Such toxicities are largely due to tissue damage sustained by chemotherapy, and strategies designed to limit such cellular damage to normal tissues may reduce therapy-related morbidity and mortality. In addition to their in vitro and in vivo anti-cancer effects, naturally occurring soy isoflavones have anti-inflammatory and anti-oxidant properties, and have been shown to reduce side effects of therapy in adult oncology clinical trials. This study will examine the effect of genistein, the major isoflavone component in soybeans and the most extensively studied of the soy isoflavones, on short-term side effects of myelosuppressive chemotherapy in pediatric cancer patients. Subjects will be randomized to receive either: a) 30 mg genistein daily throughout chemotherapy Cycles 1 and 2 and placebo during chemotherapy Cycles 3 and 4; or b) placebo daily during chemotherapy Cycles 1 and 2 and 30 mg genistein daily during chemotherapy Cycles 3 and 4. Investigators hypothesize that subjects will have fewer short-term therapy-related side effects during cycles of chemotherapy given in conjunction with genistein supplementation than cycles given with placebo.

DETAILED DESCRIPTION:
This is a multi-center, randomized, double blind, placebo-controlled crossover study to evaluate the effect of soy isoflavones on the short term untoward effects of myelosuppressive chemotherapy used to treat pediatric cancers. Newly diagnosed cancer patients aged 1-21 years will be registered to the study and informed consent will be obtained prior to any study-related procedures. Stratification will be based on length of chemotherapy cycles, between 14 day and 21 day cycles. Within strata registered subjects will be randomized 1:1 to one of two schedules:

Arm A: Subjects will receive genistein daily throughout chemotherapy cycles 1 and 2, and placebo during chemotherapy cycles 3 and 4

Arm B: Subjects will receive placebo daily throughout chemotherapy cycles 1 and 2, and genistein during chemotherapy cycles 3 and 4

Subjects will be assessed for safety and efficacy during each cycle with clinical labs, cytokine panels, and physical exams. Drug compliance will be monitored by use of a patient diary as well as monitoring of serum genistein levels. Adverse events will be monitored starting on Cycle 1 Day 1 through 30 days following the last day of protocol therapy (genistein/placebo).

ELIGIBILITY:
Inclusion Criteria

1. Newly diagnosed solid tumor or lymphoma with histological verification
2. Age 1 - 21 years at time of diagnosis
3. Karnofsky/Lanksy performance score of ≥ 50
4. Able to tolerate enteral medication administration
5. Planned chemotherapeutic regimen for a patient must meet all of the following criteria:

   * A known myelosuppressive regimen which includes at least two of the following agents: actinomycin, carboplatin, cisplatin, cyclophosphamide, daunorubicin, doxorubicin, etoposide, ifosfamide, topotecan
   * At least four consecutive cycles
   * Cycle length is either 14 or 21 days
   * Regimen must either alternate myelosuppressive chemotherapeutic agents in an X-Y-X-Y format, such that the same chemotherapy is given every other cycle (e.g. vincristine/doxorubicin/cyclophosphamide │ ifosfamide/etoposide), or repeat the same chemotherapeutic agents each cycle in an X-X-X-X format (e.g. repeated cycles of cisplatin/etoposide/bleomycin). Courses eligible for this trial may occur at any time during treatment provided that they are consecutive and follow the one of the described patterns. Non-myelosuppressive anti-neoplastic treatments will not be considered for the purposes of determining eligibility. Questions regarding whether or not a patient's chemotherapy plan meets inclusion criteria will be decided by the Study Chair.
6. Informed consent or parental permission and assent obtained prior to trial-related activities
7. Able and willing to comply with all study related procedures
8. Women of childbearing potential must agree to use adequate contraception prior to study entry and for the duration of study participation. Should a woman become pregnant or suspect she is pregnant while participating in this study, she should inform her treating physician immediately

Exclusion Criteria

1. Known allergy to soy or any soy-based food or supplement
2. Unable or unwilling to discontinue consuming prohibited soy-based food or supplements while participating in this study
3. Pre-existing neutropenia or neutrophil qualitative or quantitative disorder
4. Pre-existing cytopenia or bone marrow failure syndrome
5. History of gastric or duodenal ulcers or hyperacidity syndromes
6. History of Human Immunodeficiency Virus (HIV)
7. Has an active infection requiring systemic therapy
8. Planned treatment does not include myelosuppressive chemotherapy
9. Enrolled on a therapeutic or supportive care clinical trial within the last 30 days
10. Current acute or chronic leukemia diagnosis
11. Requires medication dosing via an enteral feeding tube that terminates in the duodenum or jejunum. (Enteral feeding tubes that terminate in the stomach are acceptable for study medication delivery.)
12. Pregnant or breastfeeding woman
13. Incarceration
14. Secondary malignancy, i.e. the cancer for which the patient is presently or will be receiving treatment may not be a malignancy related to prior cancer therapy
15. Any condition which might be worsened by estrogen, such as breast cancer, uterine cancer, ovarian cancer, endometriosis or uterine fibroids
16. Any condition, in the investigator's opinion, that would compromise patient safety or study outcomes
17. Anyone who, in the investigator's discretion, would be unwilling or unable to comply with study procedures

Ages: 1 Year to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 4 (Actual)
Dates: Start 2016-08; Primary Completion 2021-09 (Actual); Study Completion 2021-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: William C. Petersen, Jr., M.D., Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Started | 2 | 2
Completed | 2 | 2
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein | Total
Number analyzed (Participants) | 2 | 2 | 4
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 2 | 2 | 4
  Between 18 and 65 years | 0 | 0 | 0
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Full Range); unit: years] | 14 [12 to 16] | 10 [8 to 12] | 12 [8 to 16]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 2 | 2 | 4
  Male | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 0 | 0
  White | 2 | 2 | 4
  More than one race | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 2 | 2 | 4

OUTCOME MEASURES:

1. Primary Outcome: Time to Neutrophil Count Recovery Following Myelosuppressive Chemotherapy
Time Frame: From the first date study drug is taken until the last date that study drug is taken, about 8 - 12 weeks if there are no chemotherapy delays
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
days
  Genistein cycles | 13.75 (1.26) | 12.67 (2.08)
  Placebo cycles | 15.5 (1.73) | 13.5 (2.12)

2. Secondary Outcome: Serum Marker Levels of Inflammation Erythrocyte Sedimentation Rate (ESR; mm/hr) During Cycles of Chemotherapy
Time Frame: Once before treatment starts and then four more times while the study drug is being taken, an 8 - 16 week period if there are no chemotherapy delays
Measure: Mean (Standard Deviation); unit: mm/hr
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
mm/hr
  ESR, Genistein cycles | 14.67 (4.93) | 3.25 (1.5)
  ESR, Placebo cycles | 20.00 (5.29) | 2.50 (0.58)

3. Secondary Outcome: Number of Days That Participants Experience Adverse Events That Are Commonly Caused by Chemotherapy Treatment
Description: This includes hearing loss/tinnitus, motor neuropathy, oral mucositis
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: days
Groups:
- Arm A: Genistein Followed by Placebo - GENISTEIN Cycles; Arm A: Genistein Followed by Placebo - PLACEBO Cycles; Arm B: Placebo Followed by Genistein - PLACEBO Cycles: Genistein daily throughout chemotherapy cycles 1 and 2, and placebo daily during chemotherapy cycles 3 and 4
  Genistein: Estrogen-like compound (isoflavone) derived from soybeans
  Placebo: Pill that contains no medicine
- Arm B: Placebo Followed by Genistein - GENISTEIN Cycles: Placebo daily throughout chemotherapy cycles 1 and 2, and genistein daily during chemotherapy cycles 3 and 4
  Genistein: Estrogen-like compound (isoflavone) derived from soybeans
  Placebo: Pill that contains no medicine
Arm/Group | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles | Arm A: Genistein Followed by Placebo - PLACEBO Cycles | Arm B: Placebo Followed by Genistein - PLACEBO Cycles
Number analyzed (Participants) | 2 | 2 | 2 | 2
days
  Genistein Cycles | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Placebo Cycles | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

4. Secondary Outcome: Number of Participants Who Experience Adverse Events That Are Commonly Caused by Chemotherapy Treatment
Description: This includes hearing loss/tinnitus, motor neuropathy, oral mucositis
Time Frame: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles | Arm A: Genistein Followed by Placebo - PLACEBO Cycles | Arm B: Placebo Followed by Genistein - PLACEBO Cycles
Number analyzed (Participants) | 2 | 2 | 2 | 2
Participants
  Genistein Cycles | 0 | 0 | 0 | 0
  Placebo Cycles | 0 | 0 | 0 | 0

5. Secondary Outcome: Severity of Adverse Events That Are Commonly Caused by Chemotherapy Treatment Based on CTCAE Severity Criteria
Description: This includes hearing loss/tinnitus, motor neuropathy, oral mucositis
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: Events
Arm/Group | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles | Arm A: Genistein Followed by Placebo - PLACEBO Cycles | Arm B: Placebo Followed by Genistein - PLACEBO Cycles
Number analyzed (Participants) | 2 | 2 | 2 | 2
Events | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

6. Secondary Outcome: Number of Days That Participants Are Hospitalized or Have Prolonged Hospitalization Due to an Adverse Event
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: days
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
days
  Genistein cycles | 0.75 (0.5) | 0.5 (0.58)
  Placebo cycles | 0.5 (0.58) | 0.25 (0.5)

7. Secondary Outcome: Number of Days That Planned Cancer Treatment is Delayed Due to an Adverse Event
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: days
Arm/Group | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles | Arm A: Genistein Followed by Placebo - PLACEBO Cycles | Arm B: Placebo Followed by Genistein - PLACEBO Cycles
Number analyzed (Participants) | 2 | 2 | 2 | 2
days
  Genistein Cycles | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]
  Placebo Cycles | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0] | 0 [0 to 0]

8. Secondary Outcome: Percentage of Participants Requiring Reduced Treatment Doses Due to an Adverse Event
Time Frame: as for outcome 1
Measure: Number; unit: percentage of participants
Arm/Group | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles | Arm A: Genistein Followed by Placebo - PLACEBO Cycles | Arm B: Placebo Followed by Genistein - PLACEBO Cycles
Number analyzed (Participants) | 2 | 2 | 2 | 2
percentage of participants | 0 | 0 | 0 | 0

9. Secondary Outcome: Number of Days That Antimicrobial Treatment is Administered
Time Frame: as for outcome 1
Measure: Mean (Full Range); unit: days
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
days
  Genistein cycles | 0 [0 to 0] | 0 [0 to 0]
  Placebo cycles | 0 [0 to 0] | 5 [0 to 5]

10. Secondary Outcome: Number of Cycles Where Granulocyte-colony Stimulating Factor (G-CSF) is Administered
Time Frame: as for outcome 1
Measure: Number; unit: cycles
Units Other Than Participants: cycles
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
Number analyzed (cycles) | 4 | 4
cycles
  Genistein cycles | 2 | 0
  Placebo cycles | 0 | 0

11. Secondary Outcome: Number of Times That a Blood Product is Administered for Anemia, Decreased Platelets, Abnormal Bleeding, or the Subject's Best Interest
Time Frame: as for outcome 1
Measure: Mean (Standard Deviation); unit: transfusions
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
transfusions
  Genistein cycles | 0.75 (0.96) | 1.00 (1.15)
  Placebo cycles | 1.25 (0.50) | 0.75 (0.96)

12. Secondary Outcome: Serum Marker Levels of Inflammation C-reactive Protein (CRP; mg/dL) During Cycles of Chemotherapy
Time Frame: as for outcome 2
Measure: Mean (Standard Deviation); unit: mg/dL
Arm/Group | Arm A: Genistein Followed by Placebo | Arm B: Placebo Followed by Genistein
Number analyzed (Participants) | 2 | 2
mg/dL
  CRP, Genistein cycles | 0.37 (0.29) | 0.13 (0.05)
  CRP, Placebo cycles | 0.33 (0.26) | 0.15 (0.10)

ADVERSE EVENTS:
Time Frame: All AEs collected through 30 days after the last study supplement dose. In addition, investigators must report any deaths, SAEs, other AEs of concern that are believed to be related to the investigational intervention, cancer progression, cancer relapse, and secondary malignancies through six months after the end of the study intervention.
Arm/Group | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles | Arm A: Genistein Followed by Placebo - PLACEBO Cycles | Arm B: Placebo Followed by Genistein - PLACEBO Cycles
All-Cause Mortality (participants affected / at risk) | 0/2 | 1/2 | 0/2 | 0/2
Serious Adverse Events (participants affected / at risk) | 1/2 | 1/2 | 1/2 | 1/2
Other Adverse Events (participants affected / at risk) | 2/2 | 2/2 | 0/2 | 0/2
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles (N=2) | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles (N=2) | Arm A: Genistein Followed by Placebo - PLACEBO Cycles (N=2) | Arm B: Placebo Followed by Genistein - PLACEBO Cycles (N=2)
febrile neutropenia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | 1 (1) | 1 (1)
OTHER ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Arm A: Genistein Followed by Placebo - GENISTEIN Cycles (N=2) | Arm B: Placebo Followed by Genistein - GENISTEIN Cycles (N=2) | Arm A: Genistein Followed by Placebo - PLACEBO Cycles (N=2) | Arm B: Placebo Followed by Genistein - PLACEBO Cycles (N=2)
Anemia (Blood and lymphatic system disorders) | 1 (1) | 1 (1) | NA | NA
Febrile Neutropenia (Blood and lymphatic system disorders) | 1 (2) | 1 (1) | NA | NA
Abdominal pain (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Vomiting (Gastrointestinal disorders) | 1 (1) | 1 (1) | NA | NA
Nausea (Gastrointestinal disorders) | 1 (1) | 2 (2) | NA | NA
Diarrhea (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Anal mucositis (Gastrointestinal disorders) | 1 (1) | 0 (0) | NA | NA
Fatigue (General disorders) | 1 (1) | 1 (1) | NA | NA
Fever (General disorders) | 1 (1) | 1 (2) | NA | NA
Lymphocyte count decreased (Investigations) | 1 (1) | 0 (0) | NA | NA
Neutrophil count decreased (Investigations) | 2 (3) | 1 (4) | NA | NA
Platelet count decreased (Investigations) | 2 (9) | 1 (9) | NA | NA
White blood cell count decreased (Investigations) | 2 (2) | 1 (1) | NA | NA
Headache (Nervous system disorders) | 1 (3) | 1 (1) | NA | NA
Peripheral sensory Neuropathy (Nervous system disorders) | 1 (1) | 0 (0) | NA | NA
sinus tachycardia (Cardiac disorders) | 0 (0) | 1 (1) | NA | NA
Prolonged QTC interval (Cardiac disorders) | 0 (0) | 1 (4) | NA | NA
Hypotension (Vascular disorders) | 0 (0) | 1 (1) | NA | NA
Sore throat (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | NA
Cough (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 1 (1) | NA | NA
Bruising (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | NA | NA
Bladder infection (Immune system disorders) | 0 (0) | 1 (1) | NA | NA
Pain (General disorders) | 0 (0) | 1 (1) | NA | NA
Malaise (General disorders) | 0 (0) | 1 (1) | NA | NA
Methemoglobinemia (Blood and lymphatic system disorders) | 0 (0) | 1 (1) | NA | NA
Eye infection (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Sinusitis (Infections and infestations) | 0 (0) | 1 (1) | NA | NA
Upper respiratory infection (Infections and infestations) | 0 (0) | 1 (1) | NA | NA

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2017-06-30): https://cdn.clinicaltrials.gov/large-docs/88/NCT02624388/Prot_SAP_000.pdf